CLINICAL TRIAL: NCT05106023
Title: A Prospective, Single-center Clinical Study to Explore the Efficacy and Safety of SHR-1701 Combined With Temozolomide in the Treatment of Advanced Melanoma
Brief Title: To Explore the Efficacy and Safety of SHR-1701 Combined With Temozolomide in the Treatment of Advanced Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yong Chen (Other)
Responsible Party: Sponsor-Investigator, Yong Chen, Chief Physician, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM-1st-IIT-SHR1701-TMZ
Record Dates: First submitted 2021-11-01; First posted 2021-11-03 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — SHR-1701; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1701 combined with temozolomide (Experimental): SHR-1701 combined with temozolomide
  Interventions: Drug: SHR-1701; Drug: Temozolomide

INTERVENTIONS:
Drug: SHR-1701 — SHR-1701 combined with temozolomide
  Other Names: SHR1701
Drug: Temozolomide — SHR-1701 combined with temozolomide

SUMMARY:
This study is being conducted to explore the efficacy and safety of SHR-1701 combined with temozolomide in the treatment of advanced melanoma.

DETAILED DESCRIPTION:
This trial is a prospective, single-center, single-arm clinical research. Based on current experience, single agent immunotherapy has limited efficacy in advanced melanoma. SHR-1701 is a novel immunotherapy drug . Preclinical data suggest that temozolomide selectively depletes regulatory T cells. This potential immunomodulatory effect of temozolomide provides rationale for combination with SHR-1701. This study is aiming to evaluate the efficacy and safety of SHR-1701 combined with temozolomide in patients with advanced melanoma. The safety and efficacy of this study will be assessed through ORR, DCR,PFS, OS , and adverse effects as graded by CTCAE 5.0.

ELIGIBILITY:
Inclusion Criteria:

* Has unresectable Stage III or Stage IV or melanoma per American Joint Committee on Cancer (AJCC) staging system version 8. At least one measurable lesion conforming to RECIST 1.1 criteria.
* No previously received systematic therapy.
* The toxicity of prior treatment has recovered to ≤1 grade according to CTCAE 5.0.
* ECOG score 0-1.
* The expected survival time is ≥ 12 weeks.
* Adequate organ and bone marrow function.
* Female subjects of childbearing age must undergo a serum pregnancy test within 7 days before the commencement of the study and the results are negative, and are willing to use a medically approved high potency contraceptive method during the study period and within 3 months after the last administration of the study drug; For male subjects whose partner is a female of childbearing age, they should be surgically sterilized or agree to use an effective method of contraception during the study period and for 3 months after administration of the last study.
* Willing to consent and signed the informed consent, and able comply with the planned visit, research treatment, laboratory examination and other test procedures.

Exclusion Criteria:

* History of other malignant tumors, except for cured skin basal cell carcinoma, squamous cell carcinoma of skin, superficial bladder carcinoma, papillary thyroid carcinoma, intraductal carcinoma and cervical carcinoma in situ.
* Has ocular melanoma.
* The first study drug treatment was less than 4 weeks from the last systematic antitumor therapy or 5 half-lives from the last targeted therapy; less than 4 weeks from major surgery; less than7 days from immunosuppressive drug; less than 3 weeks from immunomodulatory; less than 4 weeks from live attenuated vaccine.
* Systemic antibiotic use for 7 days within 4 weeks prior to initial administration, or unexplained fever during screening/prior to initial administration.
* With active autoimmune disease or a history of autoimmune disease.
* With history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* With immunodeficiency, eg HIV, HBV, HCV.
* Have a clear history of serious and uncontrolled other disease or mental disorders.
* Has a bleeding tendency or abnormal clotting function.
* Subjects with central nervous system disease or brain metastases.
* Known to be allergic to the active ingredients or excipients in this study.
* Other situations that the researcher considers inappropriate to participate in the research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR (Objective Response Rate) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Containing the incidence of complete response (CR) and partial response (PR). Evaluated according to RECIST 1.1 criteria, subjects received their first tumor imaging evaluation at 6 weeks after the treatment start, followed by imaging evaluation every 2 cycles.

SECONDARY OUTCOMES:
PFS (Progression-Free-Survival) | From date of treatment start until the date of progression or the date of death due to any cause, assessed up to 12 months
  From date of treatment start until the date of progression or the date of death due to any cause. Evaluated according to RECIST 1.1 criteria, subjects received their first tumor imaging evaluation at 6 weeks after the treatment start, followed by imaging evaluation every 2 cycles.
DCR (Disease Control Rate) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Containing the incidence of complete response (CR), partial response (PR) and stable disease (SD).Evaluated according to RECIST 1.1 criteria, subjects received their first tumor imaging evaluation at 6 weeks after the treatment start, followed by imaging evaluation every 2 cycles.
OS (overall survival) | From date of treatment start until the date of death from any cause or censored at the last day that the subjects are documented to be alive, whichever came first, assessed up to 36 month
  From date of treatment start to any cause death or last follow-up.
6mPFS | Up to 6 months
  6-month- Progression-Free-Survival rate. Evaluated according to RECIST 1.1 criteria, subjects received their first tumor imaging evaluation at 6 weeks after the treatment start, followed by imaging evaluation every 2 cycles.
Adverse events (per CTCAE v5.0 criteria) | Up to 12months
  To evaluate the adverse events of subjects with advanced melanoma after treated with SHR-1701 plus temozolomide

CONTACTS AND LOCATIONS:
Overall Officials: yong chen, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No